CLINICAL TRIAL: NCT05936606
Title: A Randomized Comparison of TAILOReD Anti-Platelet Therapy According to Platelet Reactivity Versus Uniform Clopidogrel Monotherapy Beyond 12 Months After Drug-eluting Stent Implantation in High-risk Patients: TAILOR-DAPT
Brief Title: Tailored Anti-platelet Therapy After DES Implantation in High-risk Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2023-0175
Record Dates: First submitted 2023-05-22; First posted 2023-07-10 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; antiplatelet therapy; platelet reactivity
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to receive either standard clopidogrel monotherapy or tailored antiplatelet therapy at 12 months after DES implantation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Uniform Therapy (Active Comparator): Patients will continue clopidogrel monotherapy for 24 months from randomization, irrespective of their PRU measurement.
  Interventions: Drug: Clopidogrel monotherapy
- Tailored Therapy (Experimental): Patients in the intervention arm will receive tailored anti-platelet therapy according to PRU and bleeding risk
  Interventions: Drug: Tailored anti-platelet therapy

INTERVENTIONS:
Drug: Clopidogrel monotherapy — Patients will receive clopidogrel monotherapy (75 mg qd) for 24 months after randomization, irrespective of PRU value or bleeding risk.
  Arms: Uniform Therapy
Drug: Tailored anti-platelet therapy — In the tailored therapy arm, non-HPR (PRU<208) patients will continue clopidogrel monotherapy until the end of the study at 24 months from randomization, while HPR (PRU≥208) patients will receive dual anti-platelet therapy according to the clinical diagnosis at the time of drug-eluting stent placement: High-risk patients with prior myocardial infarction will receive ticagrelor 60 mg twice daily wiht aspirin 100 mg daily, while the remainder will receive clopidogrel 75 mg daily with aspirin 100 mg daily. For HBR patietns, early cessation of dual antiplatelet therapy or aspirin monotherapy could be considered at the investigator's discretion.
  Arms: Tailored Therapy

SUMMARY:
Clopidogrel monotherapy has been found effective in reducing ischaemic cardiovascular and haemorrhagic complications in patients with drug-eluting stent (DES) placement. However, concerns remain about the safety of long-term clopidogrel monotherapy in high-risk patients with HPR (high platelet reactivity) who do not respond adequately to clopidogrel. This study aims to evaluate the effectiveness of a patient-tailored antiplatelet therapy strategy that considers platelet aggregation in high-risk patients with DES placement beyond 12 months after stenting.

DETAILED DESCRIPTION:
This study will randomly assign eligible participants who underwent drug-eluting stent placement and have maintained the standard antiplatelet therapy for 12 months to either a control group or an intervention group. The control group will continue receiving clopidogrel monotherapy for 24 months regardless of their PRU (platelet reactivity unit) values. The intervention group will receive personalized antiplatelet therapy based on their PRU values: for non-HPR patients (PRU<208), clopidogrel monotherapy will be continued; for HPR patients (PRU≥208), dual antiplatelet therapy will be prescribed based on clinical diagnosis at the time of stent implantation and individual patients' ischemic/bleeding risk profiles. Patients (≥50 years) who presented with acute myocardial infarction at the time of coronary intervention, and have high-risk characteristics (① ≥65 years ② multi-vessel disease ③ diabetes mellitus ④ chronic kidney disease ⑤ recurrent myocardial infarction) will receive ticagrelor 60 mg twice daily with aspirin, whereas the remainder will receive clopidogrel with aspirin. For high-bleeding-risk patients with two or more major bleeding risk factors according to ARC-HBR, the investigator may consider early discontinuation of dual antiplatelet therapy or de-escalation therapy like aspirin monotherapy based on the patient's risk profile. The treatment assignment ratio is 1:1. The study period will be up to 24 months from the time of randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Patients > 18 years old
2. Patients who previously underwent percutaneous coronary intervention with drug-eluting stent implantation 12 months (± 3 months) ago.
3. At least one high risk characteristics of ischemic events

High risk patients

1. Acute coronary syndrome
2. Previous history of cerebrovascular accidents
3. Previous history of peripheral artery intervention
4. Heart failure
5. Diabetes mellitus requiring medication
6. Chronic kidney disease (regardless of requirement of renal replacement therapy)

High risk lesions

1. Left main disease
2. Multivessel disease, 2- or 3- vessels
3. Bifurcation lesions requiring 2 or more stents
4. Chronic total occlusion
5. In-stent restenosis
6. Graft lesions
7. Diffuse long lesion requiring stent(s) with total stent length ≥28 mm
8. Lesion at small sized vessel requiring stent(s) with stent diameter ≤2.5 mm
9. Calcified lesions requiring atherectomy

Exclusion Criteria:

1. Patients > 80 years old
2. Pregnant women or women with potential childbearing
3. Life expectancy < 1 year
4. Refusal or inability to understand of informed consent
5. Patients eligible to long-term anticoagulation therapy
6. Patients with major bleeding events in previous 3 months before randomization

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3434 (Estimated)
Dates: Start 2023-08-16 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Net Clinical Adverse Clinical Events (NACE) for 24 months | upto 2 years after randomization
  A composite of all-cause of death, myocardial infarction (MI), stent thrombosis, stroke, or BARC type 2, 3, or 5 bleeding

SECONDARY OUTCOMES:
All-cause death | upto 2 years after randomization
Cardiovascular death | upto 2 years after randomization
Myocardial infarction | upto 2 years after randomization
Stent thrombosis | upto 2 years after randomization
Ischemia-driven target vessel revascularization | upto 2 years after randomization
Any revascularization | upto 2 years after randomization
Stroke | upto 2 years after randomization
Bleeding Academic Research Consortium (BARC) type 2, 3, or 5 bleeding | upto 2 years after randomization
Bleeding Academic Research Consortium (BARC) type 3 or 5 bleeding | upto 2 years after randomization
Bleeding Academic Research Consortium (BARC) type 2 bleeding | upto 2 years after randomization
Bleeding Academic Research Consortium (BARC) type 3 bleeding | upto 2 years after randomization
Bleeding Academic Research Consortium (BARC) type 5 bleeding | upto 2 years after randomization
All-cause death, myocardial infarction, or stroke | upto 2 years after randomization
Cardiovascular death, myocardial infarction, stent thrombosis, or stroke | upto 2 years after randomization
All-cause death, myocardial infarction, stent thrombosis, stroke, or BARC type 3 or 5 bleeding | upto 2 years after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Byeong-Keuk Kim, Principal Investigator — Severance Cardiovascular Hospital
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No